CLINICAL TRIAL: NCT06787976
Title: Effect of Dolutegravir + Tenofovir Disoproxil Fumarato/Emtricitabina Compared With Darunavir/Cobicistat + Tenofovir Disoproxil/Fumarato /Emtricitabina on the Severity of Neuropsychiatric Effects al 12 Weeks in Antirretroviral Treatment-Naive Adults With HIV-1 Infection
Brief Title: Effect of Dolutegravir Compared With Darunavir/Cobicistat on the Severity of Neuropsychiatric Effects al 12 Weeks in Antirretroviral Treatment-Naive Adults.
Acronym: MORFEO
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Instituto Mexicano del Seguro Social (Other Government)
Responsible Party: Principal Investigator, José Antonio Mata Marín, Principal Investigator, Instituto Mexicano del Seguro Social
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: F-2024-3502-050
Record Dates: First submitted 2024-10-25; First posted 2025-01-22 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2024-08

CONDITIONS: HIV; Insomnia; Anxiety
Keywords: INSTI; HIV; Dolutegravir; Darunavir; Suicide; Depression; Anxiety
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Anxiety Disorders; Suicide; Depression | interventions — dolutegravir; Darunavir; Cobicistat

STUDY DESIGN:
Intervention Model Description: Open-label, randomized, clinical trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- DTG + TDF/FTC (Experimental): Dolutegravir + Tenofovir Disoproxil Fumarate / Emtricitabine
  Interventions: Drug: Dolutegravir (DTG)
- DRV/c + TDF/FTC (Active Comparator): Darunavir/Cobicistat + Tenofovir Disoproxil Fumarate / Emtricitabine
  Interventions: Drug: Darunavir/Cobicistat (FDC)

INTERVENTIONS:
Drug: Dolutegravir (DTG) — Dolutegravir + Tenofovir Disoproxil Fumarate / Emtricitabine
  Arms: DTG + TDF/FTC
Drug: Darunavir/Cobicistat (FDC) — Darunavir Cobicistat + TDF/FTC
  Arms: DRV/c + TDF/FTC

SUMMARY:
This clinical trial aimed at evaluating changes in neuropsychiatric scales for depression, anxiety, insomnia, and sleep quality in people living with HIV (PLHIV) who initiate antiretroviral therapy (ART) with a regimen of Dolutegravir (DTG) or Darunavir/Cobicistat (DRV/c), both combined with tenofovir disoproxil fumarate/emtricitabine (TDF/FTC).

DETAILED DESCRIPTION:
This clinical trial aims to evaluate changes in neuropsychiatric scale (NPS) scores among Mexican men living with HIV who present baseline NPS symptoms and are naïve to antiretroviral therapy (ART). Participants will initiate either a Dolutegravir (DTG)-based regimen or a Darunavir/Cobicistat (DRV/c)-based regimen, both combined with tenofovir disoproxil fumarate/emtricitabine (TDF/FTC). All patients will undergo a psychiatric evaluation prior to ART initiation. Treatment discontinuation will be considered for participants experiencing an exacerbation of NPS symptoms associated with grade ≥2 adverse events. NPS scores will be assessed and compared at weeks 4 and 12.

ELIGIBILITY:
Inclusion Criteria:

* Patients living with HIV not experienced to ART
* Age ≥ 18 years.
* eGFR >60 mL/min
* Beneficiaries of the Mexican Social Security Institute treated at the "La Raza" National Medical Center
* Patients with a baseline ISI scale score: ≥8-14 points
* Patients with a baseline PHQ-9 scale score: 5-9 points
* Patients with a baseline HADS-A scale score: 8-10 points
* Patients with a baseline HADS-D scale score: 8-10 points
* Patients with a baseline Pittsburgh scale score: 5-7 points.

Exclusion Criteria:

* Patients with use of antidepressants/anxiolytics prior to starting ART
* Any Contraindication for the use of second generation INSTI or IP ART regimen
* Coinfection with Hepatitis C Virus
* Known resistance mutations to any of the components of both treatment regimens.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2025-06-19 (Estimated); Primary Completion 2025-12-21 (Estimated); Study Completion 2026-01-25 (Estimated)

PRIMARY OUTCOMES:
Change in neuropsychiatric scales for Insomnia | 12 weeks
  Change in scales evaluating the severity of neuropsychiatric effects (Insomnia Severity Index (ISI) in patients living with HIV who are naïve to antiretroviral therapy who initiate therapy with Dolutegravir + Tenofovir Disoproxil Fumarate/Emtricitabine compared to Darunavir/cobicistat + Tenofovir Disoproxil Fumarate/Emtricitabine at 12 weeks of treatment.

SECONDARY OUTCOMES:
Discontinuation of ART due to Neuropsychiatric adverde effects | 12 weeks
  Number of patient discontinuation of ART in patients living with HIV who are naïve to antiretroviral therapy who start therapy with Dolutegravir + Tenofovir Disoproxil Fumarate/Emtricitabine compared to Darunavir/cobicistat + Tenofovir Disoproxil Fumarate/Emtricitabine after 12 weeks of treatment due to neuropsychiatric.
Risk factor associated with increase in neuropsychiatric scales | 12 weeks
  Identify the risk factors associated with the change in neuropsychiatric scales in patients living with HIV who are naïve to antiretroviral therapy and who initiate therapy with Dolutegravir + Tenofovir Disoproxil Fumarate/Emtricitabine compared to Darunavir/cobicistat + Tenofovir Disoproxil Fumarate/Emtricitabine at 12 weeks of treatment.

IPD SHARING:
Plan to Share IPD: No
Our institution does not allow us to share personal information